CLINICAL TRIAL: NCT00427557
Title: Use of Umbilical Cord Blood Cell in the Preparative Regimen of Patients With Advanced Hematologic Malignancies Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Cellular Therapy With Cord Blood Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0553
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma; Leukemia; Lymphoma
Keywords: Multiple Myeloma; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Cellular Therapy; Umbilical Cord Blood Cells; Cord Blood Transplantation; Stem Cells; Stem Cell Transplantation; Allogeneic; Hematopoietic Stem Cell Transplantation; Graft vs. Host Disease; GVD; Fludarabine; Fludarabine Phosphate; Fludara; Melphalan; Rituximab; Rituxan; Leukemia; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Leukemia; Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Graft vs Host Disease | interventions — fludarabine; fludarabine phosphate; Melphalan; Rituximab; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cellular Therapy with Cord Blood Cells (Experimental): Fludarabine 30 mg/m^2 intravenous (IV) for 4 Days + Melphalan 140 mg/m^2 IV for 1 Day + Rituximab 375 mg/m^2 IV once weekly + Cord Blood Transplantation + Stem Cell Transplantation Infusion
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: Umbilical Cord Blood; Drug: Rituximab; Other: Peripheral Blood Stem Cell Infusion

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m^2 by vein for 4 Days (Day -10 through Day -7).
  Other Names: Fludara; Fludarabine Phosphate
Drug: Melphalan — 140 mg/m^2 by vein for 1 Day (Day -7).
Procedure: Umbilical Cord Blood — 1 UCB Unit by vein on Day -5.
  Other Names: UCB
Drug: Rituximab — 375 mg/m^2 by vein once weekly (Days -7, -1, +7, +14) for 4 Weeks (if appropriate).
  Other Names: Rituxan
Other: Peripheral Blood Stem Cell Infusion — Infusion of blood stem cells on Day 0.
  Other Names: SCT; Stem Cell Transplant; Allogeneic Hematopoietic Stem Cell Transplantation; AHSCT

SUMMARY:
The goal of this clinical research study is to learn if giving umbilical cord blood along with standard stem cells after high-dose chemotherapy will improve the response to a stem cell transplant. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Cord blood is a source of blood-forming cells that can be used for transplantation. Cord blood cells are taken from the umbilical cords of women who have given birth, and who have volunteered to donate their umbilical cord. Researchers hope that using cord blood before a stem cell transplant will help to reduce the risk of graft-versus-host-disease (GVHD). GVHD occurs when donor cells attack the cells of the person receiving the transplant.

If you are found to be eligible to take part in this study, you will receive chemotherapy for 5 days. You will receive fludarabine over about 30 minutes through a needle in your vein on Days 1-4. You will receive melphalan through a needle in your vein over about 30 minutes on Day 5.

On Day 7, you will receive the cord blood cells through a needle in your vein over about 30 minutes.

On Day 12, you will receive blood stem cells through a needle in your vein over 30-60 minutes. The stem cells you receive will be from a stem cell donor whose human leukocyte antigen (HLA- proteins on cells) type matches yours.

If appropriate for the disease, you will also receive rituximab about once weekly for 4 weeks, beginning on the day you receive melphalan. Rituximab is given though a needle in your vein over 2-3 hours.

You will receive the drugs tacrolimus and methotrexate to lower the risk of GVHD. Tacrolimus will be given through a needle in your vein non-stop for 2 weeks, starting 12 hours after the stem cell transplant. After the first 2 weeks, you will continue to receive tacrolimus by mouth, for at least 3 months. You will receive methotrexate though a needle in your vein over 30 minutes, starting 1 day after the stem cell transplant, for a total of 3 doses over the first 6 days after the stem cell transplant.

You will receive the G-CSF (granulocyte-colony stimulating factor) to help you blood cell counts recover. G-CSF will be given as an injection under the skin, beginning 1 week after the stem cell transplant. You will continue to receive G-CSF once a day until your blood cell counts reach a certain high enough level.

You will need to stay in the hospital for about 4 weeks beginning on Day 1. While you are in the hospital, blood (about 2 teaspoons) will be drawn every day for routine tests.

After you leave the hospital, you will return to the hospital for visits 2-3 times a week for at least 100 days after the transplant. During these visits, you will have a physical exam and blood (about 2 teaspoons) will be drawn for routine tests.

You will be asked to come back to the clinic for follow-up visits at 3, 6, 9 and 12 months after your transplant for routine safety testing. This will include a physical exam, a bone marrow biopsy, and blood (about 2 teaspoons) will be drawn for routine testing.

You will be considered off-study after the 12-month follow-up visit.

This is an investigational study. The stem cell transplant, the umbilical cord transplant, and all drugs used on this study are FDA approved. The use of umbilical cord blood and stem cells together is investigational. Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma (MM), acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), acute lymphoblastic leukemia (ALL), non-Hodgkin's lymphoma (NHL), Hodgkin's lymphoma (HL), or chronic lymphocytic leukemia (CLL) in greater than first complete remission who are candidates for a non-ablative or reduced intensity conditioning regimen.
2. Age up to 80 years.
3. A related or unrelated donor who is HLA-matched at HLA, A, B, C, DR and DQ loci is acceptable (i.e. 10/10 matched related or unrelated donor, matched with molecular high-resolution technique per current standard for the BMT program). Donor must be willing to donate peripheral blood or bone marrow progenitor cells.
4. Available cord blood unit must contain a minimum of 1.5 * 10^7 total nucleated cells per kg, and be at least a 4/6 HLA match with patient.
5. Zubrod PS less than or equal to 2 or Lansky PS greater than or equal to 50%.
6. Left ventricular ejection fraction >40%. No uncontrolled arrhythmias or symptomatic heart disease.
7. Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC) and Diffusion Capacity (DLCO) >40%.
8. Serum creatinine <2.0 mg/dL. Serum bilirubin <3 * upper limit of normal, SGPT <4 * upper limit of normal.

Exclusion Criteria:

1. Patients with active CNS disease
2. Positive Beta HCG in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
3. Serious medical or psychiatric illness likely to interfere with participation in this clinical study, including but not limited to active uncontrolled infection, uncontrolled cardiac arrhythmia or ischemic event, or uncontrolled psychosis, major depression, or mania.
4. Evidence of chronic, active hepatitis or cirrhosis, or HIV

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 05, 2007 to November 05, 2010. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: One participant of the 31 was enrolled but did not receive treatment.
Period: Overall Study
Arm/Group | Cellular Therapy With Cord Blood Cells
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cellular Therapy With Cord Blood Cells
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment
Description: Engraftment defined as first of three (3) consecutive days with Absolute neutrophil count (ANC) equal to or more than 0.5 * 10^9/L; assessed from baseline to 100 days post-engraftment.
Time Frame: Baseline to 100 days post-engraftment
Population: Analysis per protocol.
Measure: Number; unit: participants
Groups:
- Fludarabine + Melphalan + Umbilical Cord Blood Unit: Fludarabine 30 mg/m^2 given daily for four days. Melphalan 140 mg/m^2 given for one day. Umbilical Cord Blood Unit given on one day.
Arm/Group | Fludarabine + Melphalan + Umbilical Cord Blood Unit
Number analyzed (Participants) | 30
participants | 27

ADVERSE EVENTS:
Time Frame: 10 Years and 3 Months
Arm/Group | Cellular Therapy With Cord Blood Cells
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellular Therapy With Cord Blood Cells (N=30)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)
Graft Failure (General disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ischemic Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellular Therapy With Cord Blood Cells (N=30)
Graft vs Host Disease (General disorders) | 22 (41)
Blurry Vision (Eye disorders) | 2 (2)
Delayed Engraftment (General disorders) | 2 (2)
Thrombotic Thrombocytopenia Purpura (Blood and lymphatic system disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 3 (3)
Myocarditis (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 6 (6)
Low Blood Pressure (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Hemolytic Anemia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 21 (21)
Fatigue (General disorders) | 2 (2)
Fluid Overload (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 14 (14)
Mucositis (Gastrointestinal disorders) | 21 (21)
GastrointestinaI Bleed (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 30 (30)
Elevated Creatinine (Renal and urinary disorders) | 2 (2)
Hemorrhagic Cystitis (Renal and urinary disorders) | 8 (8)
Elevated Liver Function Tests (Hepatobiliary disorders) | 12 (12)
Veno Occulusive Disease (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 22 (45)
Encephalopathy (General disorders) | 2 (2)
Headache (General disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes